CLINICAL TRIAL: NCT01390506
Title: Effect of High Dose Selenium on Inflammation and Neurological Outcome After Cardiac Arrest: A Randomized, Double Blind Placebo Controlled Phase 2a Study
Brief Title: Selenium to Improve Neurological Outcome After Cardiac Arrest
Acronym: SCPR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The company did not provide the study product
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCRP2011; 2011-001074-26 (EudraCT Number)
Record Dates: First submitted 2011-07-04; First posted 2011-07-11 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; resuscitation; neurological outcome
MeSH Terms: conditions — Heart Arrest | interventions — Selenious Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium-selenite infusion (Active Comparator): Di-sodium-selenite-pentahydrate (Na 2SeO3.5H2O) in 0,9% sodium chloride is administered intravenously at a does of 3000µg on day 0, 2000µg on day 1 and 2 and at a dose of 1000µg per day on day 3-6.
  Interventions: Drug: Sodium-selenite
- Placebo (Placebo Comparator): 0.9% sodium chloride
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium-selenite — Di-sodium-selenite-pentahydrate (Na 2SeO3.5H2O) in 0,9% sodium chloride is administered intravenously at a does of 3000µg on day 0, 2000µg on day 1 and 2 and at a dose of 1000µg per day on day 3-6.
  Other Names: selenase
  Arms: Sodium-selenite infusion
Drug: Placebo — 0,9% sodium chloride is administered intravenously
  Other Names: 0,9% sodium chloride
  Arms: Placebo

SUMMARY:
After cardiac arrest and successful resuscitation it can happen that the brain function of a patient is impaired because the brain was without oxygen for a prolonged period of time. Several strategies have been studied to improve brain function after cardiac arrest. Cooling of the patients is routinely used today. The trace element selenium has several biological functions and is important for defense mechanisms against oxidative stress, which occurs after cardiac arrest and successful resuscitation. critically ill patients have low selenium blood levels. Therefore the investigators hypothesize that giving selenium after cardiac arrest and successful resuscitation might improve brain function.

DETAILED DESCRIPTION:
When cardiopulmonary resuscitation results in the return of spontaneous circulation, intensive care is required to optimize neurological recovery. The pathophysiological reactions that follow hypoxic brain injury are complex, and the mechanisms by which ischemia causes neuronal death leading to postanoxic encephalopathy are only partly understood to date. Therapeutic hypothermia improves brain function after cardiopulmonary resuscitation. Injury however can be ongoing even after the return of spontaneous circulation, giving the clinician an additional window of opportunity to treat and protect the injured brain [5]. Therefore there is an unmet clinical need for further therapeutic strategies. Strategies to counteract the deleterious effects of oxygen-derived free radicals after cerebral reperfusion have been studied for long.

The trace element selenium is part of the enzyme glutathione peroxidase which belongs to the endogenous defence mechanisms against oxidative stress. Clinical data suggest that supplementation of selenium may be beneficial in critically ill patients and in neurodegenerative diseases including, among others, Parkinson's disease, stroke, and epilepsy, where oxidative stress plays an important pathophysiological role. In SIRS, sepsis and septic shock doses up to 4000µg per day have been proven to be safe A recent retrospective analysis supported the hypothesis that early administration of selenium may improve neurological outcome after cardiac arrest.

Therefore the purpose of this study is to explore the influence of early administration of selenium on neurological outcome after cardiopulmonary resuscitation by a randomized, placebo-controlled, single-center study.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac arrest
* Successful Resuscitation
* Age >18

Exclusion Criteria:

* Polytrauma
* Pregnancy
* Any condition that makes it likely that the patient will not survive 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
neuron specific enolase | 72 hours
  Reduction of neuron specific enolase below by more than 4.4 µg/l at 72 hours after admission to the hospital

SECONDARY OUTCOMES:
inflammation | 7 days
  Reduction of C-reactive protein, procalcitonin, interleukin 6
oxidative stress markers | 7 days
  Reduction in peroxide, peroxidase, OLAB, MDA-LDL IG, TAC, ADMA, selenium and glutathione peroxidase levels
neurological function | 6 months
  Improvement of NIH stroke scale and Glasgow Pittsburgh Performance score
Selenium blood levels | 7 days
  Increase in selenium levels in whole blood
glutathion peroxidase plasma levels | 7 days
  Improvement in glutathion peroxidase plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Stadlbauer, MD, Principal Investigator — Department of Internal Medicine, Medical University of Graz
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria